CLINICAL TRIAL: NCT06747923
Title: A Randomized, Double-blind, Placebo-controlled, Parallel, Multicenter, Exploratory Phase IIa Clinical Trial to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic Properties of SB17170 in Idiopathic Pulmonary Fibrosis (IPF) Patients.
Brief Title: SB17170 Phase 2 Trial in IPF Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SPARK Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMARTT-004
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: IPF; Idiopathic Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis (IPF)
Keywords: HMGB1
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SB17170 of A mg, Single dose (Experimental)
  Interventions: Drug: SB17170
- SB17170 of B mg, Single dose (Experimental)
  Interventions: Drug: SB17170
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB17170 — Taking SB17170 orally once a day
  Arms: SB17170 of A mg, Single dose; SB17170 of B mg, Single dose
Drug: Placebo — Taking Placebo orally once a day
  Arms: Placebo

SUMMARY:
This clinical trial is a 2:2:1 randomized, double-blind, placebo-controlled, parallel group, exploratory phase II trial. The main objective of this trial is to compare and evaluate change in FVC compared to placebo by administering SB17170 to moderate to severe patients with IPF. This clinical trial treatment involves administering SB17170 or placebo for 12 weeks.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a progressive respiratory disease characterized by a scarring process of the lung, bringing patients to respiratory failure and death in 3-5 years from diagnosis.

Subjects who meet the inclusion/exclusion criteria as a result of the screening test shall be randomized into Test Group 1 (SB17170 A mg), Test Group 2 (SB17170 B mg) and Control Group (Placebo for SB17170) in 2:2:1. Subjects who have been randomized will orally take 2 capsules once daily after a meal according to their assigned administration group for 12 weeks from the date they are prescribed the investigational product.

Safety and tolerability at 12 weeks after randomization, and efficacy at 4 & 12 weeks will be assessed. The subject who has completed 12 weeks of treatment shall visit the trial site after 1 week (Visit 7, EOS) for a follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male/female 40 years or older at the time of obtaining informed consent
2. Patients diagnosed with idiopathic pulmonary fibrosis who meet the following criteria:

   * Patients with idiopathic pulmonary fibrosis who are confirmed by chest High-Resolution Computed Tomography (HRCT) scan
   * Patients with Usual Interstitial Pneumonia (UIP) or probable UIP HRCT pattern consistent with a diagnosis of idiopathic pulmonary fibrosis confirmed through central reading of chest HRCT before the baseline visit
3. Patients with a history of idiopathic pulmonary fibrosis treatment who meet the defined criteria
4. Patients with Forced Vital Capacity (FVC) ≥ 45% of the normal predicted value at the screening visit
5. Patients meeting pulmonary function test criteria at the screening visit
6. Patients who have received the explanation of this clinical trial and voluntarily agreed and signed the informed consent form

Exclusion Criteria:

1. When there is a primary disease showing UIP patterns (rheumatoid arthritis-related interstitial lung disease, connective tissue disease-related interstitial lung disease, etc.) and/or other clinically significant lung abnormalities
2. Patients with confirmed acute exacerbation of IPF within 6 months prior to screening and/or during the screening period
3. Patients with lower respiratory tract infections requiring antibiotic treatment
4. Patients who underwent major surgery within 3 months before screening or have major surgery planned during the clinical trial
5. Patients with a history of malignancy or documented evidence of active or suspected malignancy within 5 years prior to screening
6. Patients with evidence of active infection
7. Patients with the following cardiovascular and cerebrovascular diseases at the time of screening:

   * Severe hypertension within 3 months
   * Myocardial infarction or unstable angina within 6 months
   * History of thrombotic events within 6 months
   * Diagnosis of heart failure within 6 months
8. Patients with pulmonary hypertension
9. Patients who are unable to take drugs orally or have a history of major gastrointestinal surgery or pathological findings that may affect the absorption of the investigational product
10. Patients with Human Immunodeficiency Virus (HIV) infection or active hepatitis B or C

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in FVC (ml) | Week 12
  Forced vital capacity (FVC) is the total amount of air exhaled during the lung function test.

SECONDARY OUTCOMES:
Change from baseline in FVC (%) | Week 12
  Change from baseline in FVC (%) compared to normal predicted values at 12 weeks
Change from baseline in DLCO | Week 12
  DLCO was a measurement to determine the extent to which oxygen passes from the air sacs of the lungs into the blood.
Change from baseline in quality of life and symptoms | Week 12
  Living with Pulmonary Fibrosis (L-PF) questionnaire
  : Scores range from 0 to 100, with higher numbers indicating a greater impairment.
Change from baseline in quality of life and symptoms | Week 12
  EuroQoL Five-Dimensional Instrument(EQ-5D)
  : Scores range from -0.594 to 1.0, with higher numbers indicating a better health
Change from baseline in quality of life and symptoms | Week 12
  UCSD Shortness of Breath Questionnaire
  : Scores range from 0 to 120, with higher numbers indicating greater shortness of breath.

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Myong Ji Hospital, Goyang
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Seoul Asan Hospital, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No